CLINICAL TRIAL: NCT03222492
Title: Evaluation of Brentuximab Vedotin for Diffuse Cutaneous Systemic Sclerosis BRAVOS: A Phase 1/2 Multicenter Randomized, Double Blinded, Safety Study (ITN075AI)
Brief Title: Brentuximab Vedotin for Systemic Sclerosis
Acronym: BRAVOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Seagen Inc. (Industry); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN075AI; UM1AI109565 (NIH); NIAID CRMS ID#: 38418 (Other: DAIT NIAID)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis; Scleroderma; dcSSc
Keywords: Diffuse Cutaneous Systemic Sclerosis (dcSSc); Phase 1/2 clinical trial; dose escalation randomized trial; Brentuximab vedotin
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Brentuximab Vedotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 0.6 mg/kg brentuximab vedotin (Experimental): This is the first of three ascending dose cohorts. Participants in this cohort will receive 0.6 mg/kg brentuximab vedotin (to a maximum dose 60 mg) every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Brentuximab vedotin will be administered as an intravenous infusion over 30 minutes.
  Cohort 1 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Brentuximab Vedotin
- Cohort 1: placebo (Placebo Comparator): 0.6 mg/kg placebo (to a maximum dose 60 mg). Participants in this cohort will receive 0.6 mg/kg placebo every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Placebo will be administered as an intravenous infusion over 30 minutes.
  Cohort 1 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Placebo
- Cohort 2: 1.2 mg/kg brentuximab vedotin (Experimental): This is the second of three ascending dose cohorts. Participants in this cohort will receive 1.2 mg/kg brentuximab vedotin (to a maximum dose 60 mg) every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Brentuximab vedotin will be administered as an intravenous infusion over 30 minutes.
  Cohort 2 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Brentuximab Vedotin
- Cohort 2: placebo (Placebo Comparator): 1.2 mg/kg placebo (to a maximum dose 60 mg). Participants in this cohort will receive 1.2 mg/kg placebo every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Placebo will be administered as an intravenous infusion over 30 minutes.
  Cohort 2 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Placebo
- Cohort 3: 1.8 mg/kg brentuximab vedotin (Experimental): This is the third/last of three ascending dose cohorts. Participants in this cohort will receive 1.8 mg/kg brentuximab vedotin (to a maximum dose 60 mg) every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Brentuximab vedotin will be administered as an intravenous infusion over 30 minutes.
  Cohort 3 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Brentuximab Vedotin
- Cohort 3: placebo (Placebo Comparator): 1.8 mg/kg placebo (to a maximum dose 60 mg). Participants in this cohort will receive 1.8 mg/kg placebo every 3 weeks from week 0 (initial dose) to week 21, a total of 8 treatments. Placebo will be administered as an intravenous infusion over 30 minutes.
  Cohort 3 Randomization schedule: N=6 assigned to brentuximab vedotin: N=2 assigned to placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Brentuximab Vedotin — Ascending dose cohorts. All cohorts will receive intravenous administration of study medication every 3 weeks for 21 weeks, for a total of eight doses.
  Other Names: Adcetris®
  Arms: Cohort 1: 0.6 mg/kg brentuximab vedotin; Cohort 2: 1.2 mg/kg brentuximab vedotin; Cohort 3: 1.8 mg/kg brentuximab vedotin
Biological: Placebo — Placebo control for blinding (masking), 0.95% normal saline.
  Other Names: Placebo for brentuximab vedotin
  Arms: Cohort 1: placebo; Cohort 2: placebo; Cohort 3: placebo

SUMMARY:
There is significant unmet need for effective treatment options for Diffuse Cutaneous Systemic Sclerosis (dcSSc). The present study will be a dose-escalation safety trial of brentuximab vedotin, a drug-antibody conjugate approved for the treatment of lymphoma and targeted to the protein CD30 molecule expressed on activated immune cells There is evidence for CD30 involvement in SSc. This study represents the first step in determining safety and tolerability of brentuximab vedotin in SSc.

DETAILED DESCRIPTION:
This is a multicenter prospective double blind placebo controlled dose escalation safety clinical trial with brentuximab vedotin and stable background immunosuppressive therapy in adult individuals with Diffuse Cutaneous Systemic Sclerosis (dcSSc). Adult male and female participants with dcSSc will be recruited by a collaborative group of clinical sites in the United States. Participants who meet the eligibility criteria will be enrolled without regard to gender, race, or ethnicity.

Eligible participants will be randomly assigned to study treatment, either brentuximab vedotin or placebo equivalent in a 6:2 ratio favoring brentuximab vedotin. Three dose cohorts are planned with 8 participants in each cohort, for a total of 24 participants who receive sufficient doses of the investigational medication to assess safety.

The doses planned for each ascending dose cohort include 0.6mg/kg, 1.2 mg/kg, and 1.8 mg/kg brentuximab vedotin or placebo equivalent. All cohorts will receive intravenous administration of study medication every 3 weeks for 21 weeks, for a total of eight doses. Following completion of treatment, participants will undergo follow-up visits at weeks 24, 28, 36 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Classification of Systemic Sclerosis (SSc), as defined using the 2013 American College of Rheumatology/European Union League Against Rheumatism classification of SSc;
* Diagnosis of Diffuse Cutaneous Systemic Sclerosis (dcSSc), as defined by LeRoy and Medsger, Criteria for the classification of early systemic sclerosis. J Rheumatol, 2001. 28(7): p. 1573-6;
* Disease duration ≤ 60 months (defined as time from the first non-Raynaud phenomenon manifestation);
* Modified Rodnan Skin Score (mRSS) units ≥ 15 and ≤ 45, and both of the following:

  * At least mild skin thickening (≥ 1+ mRSS) of the forearm, and
  * At least moderate skin thickening (≥ 2+ mRSS) at the planned forearm skin biopsy site.
* Documentation of at least 12 weeks of ongoing immunosuppressive therapy for SSc at the time of enrollment, and at least 4 weeks at a stable dose, of one of the following:

  * Methotrexate ≤ 25 mg/week, or
  * Mycophenolate mofetil ≤3 grams/day or mycophenolate sodium ≤2.16 grams/day, or
  * Azathioprine ≤3mg/kg/day.
* Ability to provide informed consent.

Exclusion Criteria:

* Rheumatic disease other than Diffuse Cutaneous Systemic Sclerosis (dcSSc); it is acceptable to include patients with osteoarthritis, fibromyalgia, sicca symptoms, and scleroderma-associated myopathy;
* Limited cutaneous Systemic Sclerosis (SSc) or sine scleroderma;
* Pulmonary disease with Forced Vital Capacity (FVC) ≤60% of predicted, or Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) (corrected for hemoglobin) ≤60% of predicted;
* Pulmonary hypertension (PH) or moderate to severe left ventricular dysfunction, defined as one of the following:

  * Transthoracic echocardiography demonstrating at least one of the following (unless subsequent right heart catheterization does not demonstrate PH; or unless prior right heart catheterization within one year did not demonstrate PH and echocardiography results are not significantly changed):

    * Tricuspid regurgitation jet >2.8 m/sec or estimated right ventricular systolic pressure > 42 mm Hg. or
    * At least one of the following:

      1. Abnormality of right atrial size, shape, or wall thickness consistent with PH, or
      2. Abnormality of right ventricular size, shape, or wall thickness consistent with PH, or
      3. Abnormal septal wall shape consistent with PH.
    * Left Ventricular Ejection Fraction (LVEF) <50%.
  * Right heart catheterization showing mean pulmonary artery pressure ≥25 mm Hg at rest;
  * Current use of approved medications for PH. It is acceptable to use phosphodiesterase type 5 (PDE-5) inhibitors for Raynaud's, digital ulcers, and intermittently for erectile dysfunction.
* Active scleroderma renal crisis within the 4 months prior to enrollment;
* History of moderate-to-severe lower gastrointestinal dysmotility such as current use of parenteral nutrition and/or recent history of intestinal pseudo-obstruction within 3 months prior to enrollment;
* The following medications:

  * Oral corticosteroids >10 mg/day of prednisone or equivalent within 2 weeks prior to enrollment;
  * Treatment with Intravenous Immunoglobulin (IVIG) within 12 weeks prior to enrollment;
  * Treatment with cyclophosphamide within 6 months prior to enrollment;
  * Use of investigational biologic or non-biologic medication within the past 90 days, or 5 half-lives prior to enrollment, whichever is greater;
  * Use of anti-TNF medication or other biologic medications within the past 90 days, or 5 half-lives prior to enrollment, whichever is greater;
  * Prior treatment with anti-CD20 if either of the following are true:

    * B cells ≤ lower limit of normal (LLN), or
    * Treatment with anti-CD20 has been within 12 months prior to enrollment.
  * Any prior treatment with cell-depleting therapies other than anti-CD20, including investigational agents, including but not limited to, CAMPATH(R), anti- CD4, anti-CD5, anti-CD3, anti-CD19; or
  * Any prior treatment with chlorambucil, bone marrow transplantation, or total lymphoid irradiation.
* Receipt of a live-attenuated vaccine within 3 months of study enrollment;
* Concomitant malignancies or a history of malignancy, with the exception of adequately treated basal and squamous cell carcinoma of the skin, or carcinoma in situ of the cervix;
* Major surgery (including joint surgery) within 8 weeks prior to enrollment;
* History of solid organ or hematopoietic stem cell transplantation;
* History of primary immunodeficiency;
* Comorbidities requiring systemic corticosteroid therapy, including those which have required three or more courses of systemic corticosteroids within the 12 months prior to enrollment;
* Current substance abuse or history of substance abuse within 12 months prior to enrollment;
* History of severe depression or severe psychiatric condition;
* Lack of peripheral venous access;
* Known hypersensitivity to brentuximab vedotin, a component thereof, or the excipient contained in the drug formulation;
* Severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease (or, in the investigator's opinion, any other concomitant medical condition that places the participant at risk by participating in this study), including but not limited to:

  * Uncompensated congestive heart failure (New York Heart Association Class III or VI);
  * Clinically significant active coronary artery disease (e.g., unstable angina or acute myocardial infarction within 6 months prior to enrollment);
  * Recently active cerebrovascular disease (e.g., stroke or transient ischemic attack within 6 months prior to enrollment);
  * Uncontrolled systemic hypertension;
  * Confirmed diagnosis of diabetes mellitus;
  * Pancreatitis within 30 days prior to enrollment; or
  * History or presence of peripheral neuropathy, such as mononeuritis multiplex, acute or chronic inflammatory demyelinating polyneuropathy, axonal sensorimotor neuropathies, or drug related neuropathy or neuritis.
* Evidence of infection:

  * Any infected ulcer at enrollment;
  * Active bacterial, viral, fungal, or opportunistic infections requiring systemic anti-infective therapy;
  * Evidence of current or prior infection with tuberculosis:

    * Positive QuantiFERON® - TB Gold or TB Gold Plus test results.
  * Note: Purified protein derivative (PPD) tuberculin test may be substituted for QuantiFERON® - TB Gold or TB fold Plus test.

    * Indeterminant QuantiFERON® - TB Gold test results, unless followed by a subsequent negative PPD or negative QuantiFERON® and clearance by local Infectious Disease department.
  * Evidence of current or prior infection with:

    * Human Immunodeficiency Virus (HIV), or
    * Hepatitis B Virus (as assessed by hepatitis B surface antigen, HBsAg and antibody to hepatitis B core antigen, anti-HBc), or
    * Hepatitis C Virus (HCV), with the exception of adequately treated HCV with documentation of sustained virologic response, defined as undetectable HCV RNA at least 12 weeks after the end of treatment.
  * History of progressive multifocal leukoencephalopathy (PML);
  * Hospitalization for treatment of infections, or parenteral (intravenous or intramuscular) antibacterials, antivirals, anti-fungals, or anti-parasitic agents within the past 60 days prior to enrollment;
  * Chronic infection that is currently being treated with systemic suppressive antibiotic or antiviral therapy, including but not limited to tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, and atypical mycobacteria.
  * History of significant infection or recurrent infection that, in the investigator's opinion, places the participant at risk by participating in this study.
  * Positive polymerase chain reaction (PCR) test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) within 14 days prior to enrollment.
* The following laboratory abnormalities:

  * Neutropenia (absolute neutrophil count <1500/mm^3);
  * Thrombocytopenia (platelets <100,000/mm^3);
  * Moderately severe anemia (hemoglobin, Hgb < 10 g/dL);
  * Liver function test (aspartate aminotransferase [AST], alanine aminotransferase [ALT], or alkaline phosphatase) results that are ≥ 1.5 times the upper limit of normal;
  * Serum total bilirubin > 1.5 times the upper limit of normal, or > 3 times the upper limit of normal in the presence of Gilbert's syndrome; or
  * Serum amylase and serum lipase > 1.5 times the upper limit of normal.
* Renal dysfunction, defined as either one of the following:

  * Serum creatinine > 1.5 times the upper limit of normal; or
  * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m^2.
* Pregnancy;
* Breastfeeding;
* Unwillingness to use two forms of medically acceptable contraception methods by participants and their partners (if of reproductive potential) during the study and for at least 6 months after last dose of study drug; or
* Inability to comply with study and follow-up procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, MSc, Study Chair — University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology; David Fox, MD, Study Chair — University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology
Locations (8):
- United States (8):
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - Georgetown University Medical Center: Division of Rheumatology, Washington D.C., District of Columbia
  - University of Michigan Health System: Department of Internal Medicine, Division of Rheumatology, Ann Arbor, Michigan
  - Hospital for Special Surgery, New York: Division of Rheumatology, New York, New York
  - Duke University Medical Center: Division of Rheumatology and Immunology, Durham, North Carolina
  - University of Pittsburgh Medical Center: Division of Rheumatology and Clinical, Pittsburgh, Pennsylvania
  - Medical University of South Carolina: Division of Rheumatology & Immunology, Charleston, South Carolina
  - University of Texas Houston Medical School: Division of Rheumatology and Clinical Immunogenetics, Houston, Texas

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Brentuximab Vedotin: Participants receive intravenous administration of 0.6 mg/kg Brentuximab Vedotin every 3 weeks for 21 weeks, for a total of 8 doses.
- Cohort 1 Placebo; Cohort 2 Placebo: Participants receive intravenous administration of 0.9% Normal Saline solution every 3 weeks for 21 weeks, for a total of 8 doses.
- Cohort 2 Brentuximab Vedotin: Participants receive intravenous administration of 1.2 mg/kg Brentuximab Vedotin every 3 weeks for 21 weeks, for a total of 8 doses
Period: Overall Study
Arm/Group | Cohort 1 Brentuximab Vedotin | Cohort 1 Placebo | Cohort 2 Brentuximab Vedotin | Cohort 2 Placebo
Started | 6 | 2 | 7 | 2
Completed | 6 | 2 | 5 | 2
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — COVID-19 related | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants in each cohort were randomized 6:2 to Brentuximab Vedotin or placebo, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Brentuximab Vedotin | Cohort 1 Placebo | Cohort 2 Brentuximab Vedotin | Cohort 2 Placebo | Total
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7 | 2 | 16
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (16.52) | 42.0 (22.63) | 53.1 (7.97) | 47.0 (7.07) | 49.3 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 6 | 2 | 12
  Male | 3 | 1 | 1 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 4
  Not Hispanic or Latino | 4 | 1 | 7 | 1 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 4 | 2 | 5 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 7 | 2 | 17
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.73 (5.397) | 32.49 (0.939) | 26.37 (4.831) | 22.21 (0.784) | 26.73 (4.971)
Disease Duration from Onset of Raynaud's Symptoms [Mean (Standard Deviation); unit: Months] — Raynaud's phenomenon are symptoms including localized numbness, discoloration, and sensations of cold. It is indicative of other diseases including the diffuse cutaneous form of systemic sclerosis.
  Months | 27.3 (24.05) | 45.4 (9.80) | 19.2 (7.44) | 24.7 (17.12) | 26.6 (17.35)
Disease Duration from Onset of Non-Raynaud's Symptoms [Mean (Standard Deviation); unit: Months] | 17.5 (6.70) | 46.4 (8.43) | 19.0 (8.65) | 26.2 (14.98) | 22.5 (12.18)
Baseline Modified Rodnan Skin Score (mRSS) Total Score [Mean (Standard Deviation); unit: Score] — Modified Rodnan Skin Score measures the thickness of skin. The score ranges from 0 - 3, with 0 = normal and 3 = severe. The mRSS test was performed at screening, Day 0, & at weeks 12, 24, and 48 after randomization. The baseline mRSS total score is the summation of each mRSS at these sites: right fingers, left fingers, right dorsum of hand, left dorsum of hand, right forearm, left forearm, right upper arm, left upper arm, right thigh, left thigh, right lower leg, left lower leg, right dorsum of foot, left dorsum of foot, face, anterior chest, & abdomen. The total score ranges from 0 to 51.
  Score | 31.3 (6.53) | 24.5 (2.12) | 29.0 (11.58) | 19.5 (2.12) | 28.2 (8.90)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Week 48.
Description: Adverse events were graded using the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, except for the grading of liver chemistry abnormalities. The scale ranges from grade 1 through 5, with grade 1 being the least severe and grade 5 being the most severe. Liver chemistry abnormalities were graded, from 1 through 4 (with 1 being least severe and 4 being most severe) relative to the upper limit of normal (ULN) with different grades depending on whether there was an increase in aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), or blood bilirubin.
Time Frame: Baseline through end of study (48 weeks for participants who complete the study)
Population: The safety population is defined as all participants who receive any amount of the placebo or the brentuximab vedotin study drug. Safety population is conceptually equivalent to the standard intent-to-treat population.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- 0.6 mg/kg Brentuximab Vedotin: Participants receive intravenous administration of 0.6 mg/kg Brentuximab Vedotin every 3 weeks for 21 weeks, for a total of 8 doses.
- 0.6 mg/kg Placebo; 1.2 mg/kg Placebo: Participants receive intravenous administration of 0.9% Normal Saline solution every 3 weeks for 21 weeks, for a total of 8 doses.
- 1.2 mg/kg Brentuximab Vedotin: Participants receive intravenous administration of 1.2 mg/kg Brentuximab Vedotin every 3 weeks for 21 weeks, for a total of 8 doses.
- Brentuximab Vedotin in Pooled Participants: Participants receive intravenous administration of Brentuximab Vedotin every 3 weeks for 21 weeks, for a total of 8 doses.
- Placebo in Pooled Participants: Participants receive intravenous administration of a 0.9% Normal Saline solution every 3 weeks for 21 weeks, for a total of 8 doses.
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
Proportion of participants | 0.333 [0.043 to 0.777] | 0.000 [0.000 to 0.842] | 0.571 [0.184 to 0.901] | 0.000 [0.000 to 0.842] | 0.462 [0.192 to 0.749] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 1.000, Fisher Exact — P-value is from comparing the number of participants with the AEs of interest between the two treatment groups using Fisher's exact test
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 0.444, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Week 48.
Description: as for outcome 1
Time Frame: Baseline through end of study (48 weeks)
Population: The Per Protocol 48 (PP48) is defined as the treated participants who receive at least 7 of the 8 infusions over the first 21 weeks, and who have no major protocol deviations that would affect the safety outcomes through the first 48 weeks.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.400 [0.053 to 0.853] | 0.000 [0.000 to 0.842] | 0.667 [0.094 to 0.992] | 0.000 [0.000 to 0.842] | 0.500 [0.157 to 0.843] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 0.400, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Weeks 12, 24, and 36.
Description: as for outcome 1
Time Frame: Baseline through Week 12 study visit or 12 weeks on study if the visit was missed. Baseline through Week 24 study visit or 24 weeks on study if the visit was missed. Baseline through Week 36 study visit or 36 weeks on study if the visit was missed
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
proportion of participants
  Week 12 | 0.167 [0.004 to 0.641] | 0.000 [0.000 to 0.842] | 0.143 [0.004 to 0.579] | 0.000 [0.000 to 0.842] | 0.154 [0.019 to 0.454] | 0.000 [0.000 to 0.602]
  Week 24 | 0.333 [0.043 to 0.777] | 0.000 [0.000 to 0.842] | 0.286 [0.037 to 0.710] | 0.000 [0.000 to 0.842] | 0.308 [0.091 to 0.614] | 0.000 [0.000 to 0.602]
  Week 36 | 0.333 [0.043 to 0.777] | 0.000 [0.000 to 0.842] | 0.429 [0.099 to 0.816] | 0.000 [0.000 to 0.842] | 0.385 [0.139 to 0.684] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 0.500, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Week12
Description: as for outcome 1
Time Frame: Baseline through Week 12 study visit or 12 weeks on study if the visit was missed.
Population: The Per Protocol 12 (PP12) is defined as the treated participants who receive at least 4 of the 5 infusions over the first 12 weeks, and who have no major protocol deviations that would affect the safety outcomes through the first 12 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 5 | 2 | 10 | 4
proportion of participants | 0.200 [0.005 to 0.716] | 0.000 [0.000 to 0.842] | 0.200 [0.005 to 0.716] | 0.000 [0.000 to 0.842] | 0.200 [0.025 to 0.556] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Weeks 24.
Description: as for outcome 1
Time Frame: Baseline through Week 24 study visit or 24 weeks on study if the visit was missed.
Population: The Per Protocol 24 (PP24) is defined as the treated participants who receive at least 7 of the 8 infusions over the first 21 weeks, and who have no major protocol deviations that would affect the safety outcomes through the first 24 weeks.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 4 | 2 | 9 | 4
proportion of participants | 0.400 [0.053 to 0.853] | 0.000 [0.000 to 0.842] | 0.500 [0.068 to 0.932] | 0.000 [0.000 to 0.842] | 0.444 [0.137 to 0.788] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 0.467, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 3 or Higher Adverse Event at or Before Weeks 36.
Description: as for outcome 1
Time Frame: Baseline through Week 36 study visit or 36 weeks on study if the visit was missed.
Population: The Per Protocol 36 (PP36) is defined as the treated participants who receive at least 7 of the 8 infusions over the first 21 weeks, and who have no major protocol deviations that would affect the safety outcomes through the first 36 weeks.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.400 [0.053 to 0.853] | 0.000 [0.000 to 0.842] | 0.667 [0.094 to 0.992] | 0.000 [0.000 to 0.842] | 0.500 [0.157 to 0.843] | 0.00 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 0.400, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 2 or Higher Adverse Event at or Before Weeks 12, 24, 36, and 48.
Description: as for outcome 1
Time Frame: Baseline thru Week 12 visit or 12 weeks on study if visit was missed/thru Week 24 visit or 24 weeks on study if visit was missed/thru Week 36 visit or 36 weeks on study if visit was missed/thru Week 48 visit or 48 weeks on study if visit was missed
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
proportion of participants
  Week 12 | 0.833 [0.359 to 0.996] | 0.500 [0.013 to 0.987] | 0.429 [0.099 to 0.816] | 0.000 [0.000 to 0.842] | 0.615 [0.316 to 0.861] | 0.250 [0.006 to 0.806]
  Week 24 | 1.000 [0.541 to 1.000] | 0.500 [0.013 to 0.987] | 0.714 [0.290 to 0.963] | 0.000 [0.000 to 0.842] | 0.846 [0.546 to 0.981] | 0.250 [0.006 to 0.806]
  Week 36 | 1.000 [0.541 to 1.000] | 1.000 [0.158 to 1.000] | 0.857 [0.421 to 0.996] | 0.000 [0.000 to 0.842] | 0.923 [0.640 to 0.998] | 0.500 [0.068 to 0.932]
  Week 48 | 1.000 [0.541 to 1.000] | 1.000 [0.158 to 1.000] | 0.857 [0.421 to 0.996] | 0.000 [0.000 to 0.842] | 0.923 [0.640 to 0.998] | 0.500 [0.068 to 0.932]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 0.464, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 0.500, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 0.250, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 0.167, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 0.083, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 0.083, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 2 or Higher Adverse Event at or Before Weeks 12
Description: as for outcome 1
Time Frame: Baseline through the Week 12 study visit or 12 weeks on study if the visit was missed
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 5 | 2 | 10 | 4
proportion of participants | 0.800 [0.284 to 0.995] | 0.500 [0.013 to 0.987] | 0.600 [0.147 to 0.947] | 0.000 [0.000 to 0.842] | 0.700 [0.348 to 0.933] | 0.250 [0.006 to 0.806]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 12; Test type: Superiority; p = 0.429, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 2 or Higher Adverse Event at or Before Weeks 24.
Description: as for outcome 1
Time Frame: Baseline through the Week 24 study visit or 24 weeks on study if the visit was missed.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 4 | 2 | 9 | 4
proportion of participants | 1.000 [0.478 to 1.000] | 0.500 [0.013 to 0.987] | 1.000 [0.398 to 1.000] | 0.000 [0.000 to 0.842] | 1.000 [0.664 to 1.000] | 0.250 [0.006 to 0.806]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 0.286, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 24; Test type: Superiority; p = 0.067, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 2 or Higher Adverse Event at or Before Weeks 36.
Description: as for outcome 1
Time Frame: Baseline through the Week 36 study visit or 36 weeks on study if the visit was missed.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 1.000 [0.478 to 1.000] | 1.000 [0.158 to 1.000] | 1.000 [0.292 to 1.000] | 0.000 [0.000 to 0.842] | 1.000 [0.631 to 1.000] | 0.500 [0.068 to 0.932]
Statistical Analysis 1: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 36; Test type: Superiority; p = 0.100, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Proportion of Participants That Experience at Least One Grade 2 or Higher Adverse Event at or Before Weeks 48.
Description: as for outcome 1
Time Frame: Baseline through the Week 48 study visit or 48 weeks on study if the visit was missed.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 1.000 [0.478 to 1.000] | 1.000 [0.158 to 1.000] | 1.000 [0.292 to 1.000] | 0.000 [0.000 to 0.842] | 1.000 [0.631 to 1.000] | 0.500 [0.068 to 0.932]
Statistical Analysis 1: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 0.100, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Peripheral Neuropathy at or Before Weeks 12, 24, 36, and 48.
Description: Adverse events were graded using the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, except for the grading of liver chemistry abnormalities. The scale ranges from grade 1 through 5, with grade 1 being the least severe and grade 5 being the most severe.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
proportion of participants
  Week 12 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 24 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 36 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 48 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]

13. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Peripheral Neuropathy at or Before Weeks 12
Description: as for outcome 12
Time Frame: Baseline through the Week 12 study visit or 12 weeks on study if the visit was missed.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 5 | 2 | 10 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.308] | 0.0 [0.000 to 0.602]

14. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Peripheral Neuropathy at or Before Weeks 24.
Description: as for outcome 12
Time Frame: Baseline through the Week 24 study visit or 24 weeks on study if the visit was missed.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 4 | 2 | 9 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.602] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.336] | 0.0 [0.000 to 0.602]

15. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Peripheral Neuropathy at or Before Weeks 36.
Description: as for outcome 12
Time Frame: Baseline through the Week 36 study visit or 36 weeks on study if the visit was missed.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.708] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.369] | 0.0 [0.000 to 0.602]

16. Secondary Outcome: Proportion of Participants With Grade 2 or Higher Peripheral Neuropathy at or Before Weeks 48.
Description: as for outcome 12
Time Frame: Baseline through the Week 48 study visit or 48 weeks on study if the visit was missed.
Population: 5 The Per Protocol 48 (PP48) is defined as the treated participants who receive at least 7 of the 8 infusions over the first 21 weeks, and who have no major protocol deviations that would affect the safety outcomes through the first 48 weeks.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.708] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.369] | 0.0 [0.000 to 0.602]

17. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Neutropenia at or Before Weeks 12, 24, 36, and 48.
Description: as for outcome 12
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
proportion of participants
  Week 12 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 24 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 36 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]
  Week 48 | 0.0 [0.000 to 0.459] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.410] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.247] | 0.0 [0.000 to 0.602]

18. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Neutropenia at or Before Weeks 12
Description: as for outcome 12
Time Frame: Baseline through the Week 12 study visit or 12 weeks on study if the visit was missed.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 5 | 2 | 10 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.308] | 0.0 [0.000 to 0.602]

19. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Neutropenia at or Before Weeks 24.
Description: as for outcome 12
Time Frame: Baseline through the Week 24 study visit or 24 weeks on study if the visit was missed.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 4 | 2 | 9 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.602] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.336] | 0.0 [0.000 to 0.602]

20. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Neutropenia at or Before Weeks 36.
Description: as for outcome 12
Time Frame: Baseline through the Week 36 study visit or 36 weeks on study if the visit was missed.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.708] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.369] | 0.0 [0.000 to 0.602]

21. Secondary Outcome: Proportion of Participants With Grade 3 or Higher Neutropenia at or Before Weeks 48.
Description: as for outcome 12
Time Frame: Baseline through the Week 48 study visit or 48 weeks on study if the visit was missed.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.0 [0.000 to 0.522] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.708] | 0.0 [0.000 to 0.842] | 0.0 [0.000 to 0.369] | 0.0 [0.000 to 0.602]

22. Secondary Outcome: Proportion of Participants With Any of the Following Grade 3 or Higher AEs at or Before Week 48: Peripheral Neuropathy, Neutropenia, Infectious Adverse Events, Infusions Reactions, or Progressive Multifocal Leukoencephalopathy.
Description: as for outcome 1
Time Frame: Baseline through the Week 48 study visit or 48 weeks on study if the visit was missed.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 6 | 2 | 7 | 2 | 13 | 4
proportion of participants | 0.167 [0.004 to 0.641] | 0.000 [0.000 to 0.842] | 0.143 [0.004 to 0.579] | 0.000 [0.000 to 0.842] | 0.154 [0.019 to 0.454] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

23. Secondary Outcome: Proportion of Participants With Any of the Following Grade 3 or Higher AEs at or Before Week 48: Peripheral Neuropathy, Neutropenia, Infectious Adverse Events, Infusions Reactions, or Progressive Multifocal Leukoencephalopathy.
Description: as for outcome 1
Time Frame: Baseline through the Week 48 study visit or 48 weeks on study if the visit was missed.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
Number analyzed (Participants) | 5 | 2 | 3 | 2 | 8 | 4
proportion of participants | 0.200 [0.005 to 0.716] | 0.000 [0.000 to 0.842] | 0.333 [0.008 to 0.906] | 0.000 [0.000 to 0.842] | 0.250 [0.032 to 0.651] | 0.000 [0.000 to 0.602]
Statistical Analysis 1: Comparison: 0.6 mg/kg Brentuximab Vedotin vs 0.6 mg/kg Placebo; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 1.2 mg/kg Brentuximab Vedotin vs 1.2 mg/kg Placebo; Treatment start to Week 48; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a participant signed informed consent until study completion (week 48) or until 30 days after a participant withdrew early from the study.
Groups:
- 0.6 mg/kg Placebo: Participants receive intravenous administration of 0.6 mg/kg of a 0.9% Normal Saline solution every 3 weeks for 21 weeks, for a total of 8 doses.
- 1.2 mg/kg Placebo: Participants receive intravenous administration of 1.2 mg/kg of a 0.9% Normal Saline solution every 3 weeks for 21 weeks, for a total of 8 doses.
Arm/Group | 0.6 mg/kg Brentuximab Vedotin | 0.6 mg/kg Placebo | 1.2 mg/kg Brentuximab Vedotin | 1.2 mg/kg Placebo | Brentuximab Vedotin in Pooled Participants | Placebo in Pooled Participants
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/7 | 0/2 | 0/13 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 2/7 | 0/2 | 3/13 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 6/7 | 0/2 | 12/13 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg/kg Brentuximab Vedotin (N=6) | 0.6 mg/kg Placebo (N=2) | 1.2 mg/kg Brentuximab Vedotin (N=7) | 1.2 mg/kg Placebo (N=2) | Brentuximab Vedotin in Pooled Participants (N=13) | Placebo in Pooled Participants (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg/kg Brentuximab Vedotin (N=6) | 0.6 mg/kg Placebo (N=2) | 1.2 mg/kg Brentuximab Vedotin (N=7) | 1.2 mg/kg Placebo (N=2) | Brentuximab Vedotin in Pooled Participants (N=13) | Placebo in Pooled Participants (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Forced vital capacity decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung diffusion test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to slow enrollment the study was stopped before fully enrolling cohort 2 (1.2 mg/kg) and before starting cohort 3 (1.8 mg/kg).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03222492/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT03222492/SAP_002.pdf
  • Informed Consent Form (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03222492/ICF_000.pdf